CLINICAL TRIAL: NCT02744638
Title: Double-blind, Randomized, Controlled Trial to Evaluate the Effect of a Yoghurt Containing Four Probiotic Lactobacillus Strains (L. Crispatus, L. Gasseri, L. Rhamnosus, L. Jensenii) on Bacterial Vaginosis (BV) in Adult Women
Brief Title: Effect of a Yoghurt Containing Four Probiotic Lactobacillus Strains on Bacterial Vaginosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Center Kiel GmbH (Other)
Collaborators: Dairyfem R&D GmbH (Unknown); University of Natural Resources and Life Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: DF-WCT-2014
Record Dates: First submitted 2016-03-31; First posted 2016-04-20 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-04

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; probiotics; Amsel Score; Nugent Score
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — calcium D-pantothenate, L-cysteine drug combination; Benchmarking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotic yoghurt & Arilin (Experimental): probiotic yoghurt, 2 units (125 g), containing living strains of L.crispatus, L.gasseri, L.rhamnosus, L.jensenii, each in a concentration of 1 x 107 CFU/ml product for 4 weeks Two yoghurts are consumed every day for 28 days. 2 tablets Metronidazol 500mg daily for 7 days
  Interventions: Other: probiotic yoghurt; Drug: Arilin
- chemically acidified milk & Arilin (Placebo Comparator): chemically (H3PO4) acidified milk (125g) without bacterial strains. Two products are consumed every day for 28 days. 2 tablets Metronidazol 500mg daily for 7 days
  Interventions: Other: chemically acidified milk; Drug: Arilin

INTERVENTIONS:
Other: probiotic yoghurt — verum is a liquid probiotic yoghurt containing all four probiotics as described in the arm description. Study participants consume daily two bottles (125g) during an intervention period of four weeks.
  Other Names: verum
  Arms: probiotic yoghurt & Arilin
Other: chemically acidified milk — Placebo is chemically acidified milk without bacterial strains. Study participants consume daily two bottles (125g) during an intervention period of four weeks (randomly assigned).
  Other Names: placebo
  Arms: chemically acidified milk & Arilin
Drug: Arilin — 2 tablets Arilin 500mg for 7 days
  Other Names: Metronidazol

SUMMARY:
The aim of this study is, to investigate, whether the consumption of a probiotic yoghurt containing 4 probiotic strains naturally colonizing the vagina (L. crispatus, L. gasseri, L. rhamnosus, L. jensenii) has an influence on the comfort of adult women with BV after and 3 weeks following a standard antibiotic treatment with metronidazole.

DETAILED DESCRIPTION:
Female volunteers aged ≥18 years with stable menstrual cycle or postmenopausal women presenting with a newly diagnosed bacterial vaginosis based on Amsel criteria, complying with a standard oral antibiotic treatment (Metronidazol (Arilin®) 7 days 2x500mg), willing to consume for 4 weeks the study product two times daily, complying with the dietary restrictions (s. a.) and complying with the other inclusion and exclusion criteria will be enrolled in the study. After enrollment subjects will be randomly and evenly assigned to one of the two test groups verum and placebo.The study population will be recruited in a screening examination (G1) by gynaecologists from Kiel area. This screening examination (routine examination) by gynaecologist is used to provide the diagnosis BV. After enrolment subjects will be randomly assigned to one of the two test groups verum (n=108) and placebo (n=108).

ELIGIBILITY:
Inclusion Criteria:

To be enrolled, the following criteria have to be fulfilled:

1. Woman aged ≥ 18 years with stable menstrual cycle or postmenopausal women
2. Newly diagnosed bacterial vaginosis based on Amsel criteria
3. Complies with a standard oral antibiotic treatment with Metronidazol for 7 days, 2 x 500mg/day)
4. Willing to consume for 4 weeks the study product two times daily
5. Willingness to abstain from food and supplements containing probiotics, prebiotics and other fermented products as well as dietary supplements
6. Not in menses at the time of the first examination at the gynaecologist (G1)
7. Written informed consent

Exclusion Criteria:

1. Subjects currently enrolled in another clinical study.
2. Subjects having finished another clinical study within the last 4 weeks before inclusion.
3. Infection caused by Chlamydia trachomatis
4. Infection caused by Neisseria gonorrhoea
5. Infection caused by Trichomonas vaginalis
6. Infection caused by Candida albicans or other mycosis
7. Leucocytes present in the vaginal smear
8. PAP-testing ≥ 3 (anamnestically)
9. Vulvovaginal inflammation as macroscopically identified by the gynaecologist
10. Dyspareunia
11. Pregnancy and breastfeeding
12. Chemically based contraceptives (e.g. suppositories, salves, foam, gel)
13. Irregular cycles (e.g. polymenorrhoea, metrorrhagia)
14. Dysuria
15. Infection of the urinary tract
16. Chronic or sporadic abdominal pain with exception of dysmenorrhoea
17. Any ano-rectal infection, disease, surgery in the medical history or current
18. Anus praeter
19. Hypersensitivity, allergy or idiosyncratic reaction to metronidazole or any similar active substances.
20. Hypersensitivity, allergy or idiosyncratic reaction to any component of the yoghurt (e.g. lactose intolerance, allergy against milk protein)
21. Any disease or condition which might compromise significantly the hematopoietic, renal, endocrine, pulmonary, hepatic, gastrointestinal, cardiovascular, immunological, central nervous, dermatological or any other body system with the exception of the conditions defined by the inclusion criteria.
22. History of hepatitis B and C
23. History of HIV infection
24. Regular medical treatment including OTC, which may have impact on the study aims (e.g. probiotics, antibiotic drugs, laxatives etc.)
25. Major cognitive or psychiatric disorders
26. Subjects who are scheduled to undergo hospitalization during the study period
27. Eating disorders (e.g. anorexia, bulimia) or special diets (e.g. vegan, vegetarian)
28. Present drug abuse or alcoholism, reformed alcoholic
29. Legal incapacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Rate of BV-free woman | 4 weeks
  The rate of BV-free women at the end of the yoghurt consumption period (day 28) as assessed by Nugent score

SECONDARY OUTCOMES:
Alteration (G2 - G1) of Nugent Score | 4 weeks
Alteration (G2 - G1) of symptom score based on Amsel criteria (Yes=1; No=0) and 3 (Yes=1; No=0) resulting in a score ranging from 0 to 2 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Laue, Dr. med., Principal Investigator — CRC Clinical Research Center Kiel
Locations (1):
- CRC Clinical Research Center Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No